CLINICAL TRIAL: NCT02332148
Title: A Double-blind, Placebo-controlled, Randomized Study to Assess the Safety and Efficacy of 3VM1001 Cream for the Treatment of Chronic Pain Caused by Osteoarthritis of the Knee: A Proof of Concept Study
Brief Title: Assessment of the Safety and Efficacy of 3VM1001 Cream for Treatment of Chronic Pain Caused by Knee Osteoarthritis.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CDA Research Group, Inc. (Industry)
Collaborators: 3VM Research Group, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3VM0115
Record Dates: First submitted 2015-01-05; First posted 2015-01-06 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-08

CONDITIONS: Osteoarthritis of Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 3Vm1001 (Experimental): 3VM1001 topical cream containing 10 mg/day of copper, for 30 days
  Interventions: Drug: 3VM1001
- Placebo (Placebo Comparator): Placebo for 3VM1001, topical cream without 3VM1001
  Interventions: Drug: Placebo for 3VM1001

INTERVENTIONS:
Drug: 3VM1001 — 3VM1001 topical cream for treatment of osteoarthritis of the knee
  Arms: 3Vm1001
Drug: Placebo for 3VM1001 — Topical cream placebo for 3VM1001; cream without 3VM1001
  Arms: Placebo

SUMMARY:
3VM1001 is a topical cream that may be useful for the treatment of chronic osteoarthritis of the knee. This proof of concept study is a randomized, placebo-controlled, double-blind study to compare treatment with 3VM1001 cream to an inactive cream placebo. Subjects will self-treat for 30 days.

DETAILED DESCRIPTION:
3VM1001 is a topical cream that may be useful for the treatment of chronic osteoarthritis of the knee. This proof of concept study is a randomized, placebo-controlled, double-blind study to compare treatment with 3VM1001 cream to an inactive cream placebo. Subjects will self-treat for 30 days with investigational drug or placebo. Rescue medication with acetaminophen, up to 2g daily, is permitted. This study is intended to evaluate the safety and efficacy of 3VM1001 topical cream, a copper-containing cream. Subjects will self treat with drug or placebo three times daily for 30 days. All subjects will have a total of three visits to the clinic and will complete a daily diary each day for the 30 days of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis of the knee according to American College of Rheumatology clinical radiological criteria;
* OA of knee ≥ 6 months prior to screening;
* age 40 years or older;
* subjects of childbearing potential and their partners must use effective contraception;
* women of childbearing age must have a negative pregnancy test or screening or be using an acceptable form of birth control;
* moderate to severe chronic OA pain defined as POM score between 40 mm and 90 mm;
* baseline WOMAC pain subscale score ≥ 9;
* no change in physical activity and/or therapy for the past 3 months;- all concurrent medications taken for any reason stable for 14 days;
* ability to follow protocol with reference to cognitive and situational factors (eg. stable housing, ability to attend visits;
* ability to read and write English;
* ability to apply cream without assistance;
* able to provide written informed consent.

Exclusion Criteria:

* Presence of significant medical disorder that would compromise the participant's safety to take part in the trial (e.g. cancer, immunosuppressed) or evidence of alcohol or substance abuse;
* Wilson's disease or other disorder of copper metabolism
* BMI >35
* Known hypersensitivity or allergy to any component of the product, or to acetaminophen
* Pregnant and breastfeeding women
* Transcutaneous electrical nerve stimulation and use of crutches, walkers, or wheel chairs should be excluded prior to and during treatment
* Active conditions over the area to be treated such as eczema or psoriasis, compromised integrity of the intact, superficial skin layer over the area to be treated.
* Pain in any joint other than the index joint that could interfere with the patient's assessment of pain in the index joint
* Recent injury (traumatic or sports related) to either knee causing pain and interference with daily activities (e.g. walking)
* Recent surgery/procedure to either knee causing pain that could interfere with study assessments of pain, function, and QoL.
* Extreme pain in the target knee characterized by POM score of >90 mm
* Mild pain in the target knee, characterized by POM score of < 40 mm
* Open surgery of the target knee within the last year
* Arthroscopic surgery of the target knee within the last 3 months
* Use of prohibited concomitant medications/therapies during the 30-day treatment period including:

  1. devices or therapeutic treatments for knee pain or ambulation
  2. analgesics other than acetaminophen
  3. Systemic corticosteroids
  4. other investigational drugs
  5. chemotherapeutic drugs
  6. immunotherapy
  7. topical products applied to the target knee

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-02; Primary Completion 2015-10 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Time-averaged change in pain from baseline in a standard visual analog scale | baseline and 30 days